CLINICAL TRIAL: NCT07145697
Title: The Electroencephalographic Mechanisms of Anesthesia and Human Consciousness
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, Clinical Professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Mechanisms of Consciousness
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Consciousness, Level Altered
MeSH Terms: conditions — Consciousness Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep (No Intervention): Recordering electroencephalograms during nighttime natural sleep.
- Dexmedetomidine (Experimental): Escalating concentrations until loss of responsiveness
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Escalating concentrations until loss of responsiveness
  Arms: Dexmedetomidine

SUMMARY:
In the field of general anesthesia research, the neural mechanism underlying the loss of consciousness has long been a highly core issue. It remains unclear what consciousness is and how it emerges from brain activity. By studying anesthesia and sleep, the investigators aim to reveal what happens in the brain when consciousness is lost and when it returns.

Dexmedetomidine, a widely used drug in clinical anesthetic practice, plays an important role in the anesthetic process due to its unique pharmacological properties. It hardly causes respiratory depression during the sedative and hypnotic process, which makes it occupy an important position in clinical anesthetic regimens.

The emergence of stereoelectroencephalography (SEEG) technology has brought new opportunities for research on anesthesia mechanisms. Compared with traditional electroencephalographic (EEG), SEEG can directly penetrate into deep brain structures to record electrical activities, enabling precise localization of brain regions closely related to consciousness regulation.

At present, although there have been some studies on the effects of dexmedetomidine on EEG activities, there are still many deficiencies. Most studies have focused on simple spectral analysis of EEG signals or observations of limited brain regions, lacking comprehensive multi-dimensional research on functional connectivity between brain regions, microstates, and complexity. Through monitoring key brain regions, the SEEG technology can obtain more targeted and accurate information, thereby providing strong support for comprehensively revealing the neural mechanisms of dexmedetomidine-induced loss of consciousness.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 1 - 65 years old
2. BMI: 18.5 - 25.0 kg/m²
3. ASA physical status classification: I - III
4. Patients diagnosed with drug - refractory epilepsy who, after long - term monitoring of epileptic seizures, require stereo-electroencephalography (SEEG) electrode implantation based on the clinical need for monitoring their epilepsy.
5. Patients voluntarily participate in this study and sign a written informed consent form.

Exclusion Criteria:

1. Patients with severe arrhythmia or other organic heart diseases;
2. Patients with comorbid obstructive sleep apnea-hypopnea syndrome (OSAHS);
3. Patients with hepatic or renal dysfunction; those with a history of immunodeficiency diseases , or a history of cancer/malignant tumors, or a history of autoimmune diseases, or severe cardiovascular and cerebrovascular diseases, or other diseases that may significantly reduce life expectancy;
4. Patients with any history of diseases that may affect protocol compliance (such as severe mental disorders, disturbance of consciousness; cognitive dysfunction, drug abuse or addiction, etc.);
5. Pregnant or lactating women, or those of childbearing potential who are unwilling/unable to take effective contraceptive measures;
6. Patients with known allergies to the ingredients contained in the drugs used in this study;
7. Patients who have participated in any drug clinical trial within 6 months before the screening examination;
8. Patients who are deemed unsuitable to participate in this study by the researcher.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Stereo-electroencephalography | After the patient has completed the monitoring of epileptic seizures due to clinical needs, they can participate in this test. Through test completion, an average of 3 hours.

SECONDARY OUTCOMES:
Functional connectivity | through test completion, an average of 3 hours
  permutation mutual information (PMI); stereo-electroencephalography assessment parameter
The complexity | through test completion, an average of 3 hours
  examined by permutation entropy (PE); stereo-electroencephalography assessment parameter
Phase-amplitude coupling (PAC) | through test completion, an average of3 hours.
  PAC is used to illuminate cross-frequency coordination in neurophysiological activity of electroencephalogram. stereo-electroencephalography assessment parameter
Directional connectivity | through test completion, an average of 3 hours
  symbolic conditional mutual information (SCMI) and directionality index (DI); stereo-electroencephalography assessment parameter

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital of southern theater command, PLA, Guangzhou, Guangdong, China